CLINICAL TRIAL: NCT06227208
Title: The Impact of Postoperative Opioids on Duration and Severity of Desaturation and Bradypnea in Opioid-naïve and Chronic Opioid Patients, Assessed by Continuous Vital Sign Monitoring.
Brief Title: Postoperative Opioid and Respiratory Depression in Opioid Naive and Chronic Opioid Patients
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Eske Kvanner Aasvang, Professor, head of research, MD, DmSci, Rigshospitalet, Denmark
Other Study IDs: WARD-postoperative-opioid
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Medical Complication
Keywords: Opioid-induced respiratory depression; Postoperative opioid; Opioid-naïve patients; Chronic opioid patients; Desaturation; Bradypnea; Continuous monitoring; Patient safety
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Opioid-naive patients: Opioid-naive patients are defined as the absence of any documented opioid use in the available preoperatively medical records, and are receiving opioids postoperatively
  Interventions: Device: Continuous vital sign monitoring
- Chronic opioid patients: Chronic opioid patients were defined as current or previous use of the following medications, re-gardless of the duration of use: morphine, tramadol, tapentadol, fentanyl, oxycodone, ketobe-midone, methadone, or buprenorphine. This was verified through patients' preoperative medical records. All chronic opioid users received postoperative opioids.
  Interventions: Device: Continuous vital sign monitoring
- Control group: Patients who did not receive pre- or postoperative opioids were served as the overall control group.
  Interventions: Device: Continuous vital sign monitoring

INTERVENTIONS:
Device: Continuous vital sign monitoring — Wireless monitoring system that provided continuous, non-invasive collection of their vital signs, including peripheral oxygen saturation (SpO2) and respiratory rate (RR), for up to 92 hours following surgery or until discharge. The respiratory rate was monitored via FDA-approved Isansys Lifetouch electrocardiogram (ECG) patch, which was placed on the left side of the chest. SpO2 levels were continuously recorded using the Nonin WristOx 3150, a wrist-mounted finger oximeter.

SUMMARY:
Aim: To describe the duration of desaturation and bradypnea in postoperative opioid-naïve and chronic opioid patients. Patients: 691 patients included from two previous WARD (Wireless Assessment of Respiratory and circulatory Distress) projects. Outcome: Respiratory deviations four hours after opioid administration

DETAILED DESCRIPTION:
Aim: To describe the duration of desaturation and bradypnea in postoperative opioid-naïve and chronic opioid patients within the first four hours following opioid administration in addition to the chronic dose, using a continuously wireless monitoring system.

Patients: 691 patients included from two previous WARD (Wireless Assessment of Respiratory and circulatory Distress) projects. Continuous wireless monitoring data of peripheral tissue oxygenation (SpO2) and respiratory rate (RR) was conducted in postoperative patients. Data were stratified into opioid-naïve and chronic opioid patients, based on their preoperative opioid history. Patients who did not receive opioids postoperatively were served as the control group. Data was evaluated one hour before and four hours after opioid administration. The primary outcome was the cumulative duration of SpO2 <88%.

ELIGIBILITY:
Inclusion Criteria:

* Patients from studies WARD Surgery Observational [gov: NCT03491137]
* The control group from WARD Surgery Randomized Controlled Trial [gov: NCT04640415]

Exclusion Criteria:

* Less than 30 minutes of continuous monitoring data within the 60-minute window prior to opioid administration
* Less than 120 minutes (<50% of theoretical maximum) of monitoring data available during the four-hour observation period
* Patients who received transdermal fentanyl as postoperative opioid
* Patients with a baseline saturation or respiratory rate below the prespecified thresholds
* Patients with a BMI of ≥40 or diagnosed with COPD were excluded in the analysis of SpO2 <92%

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients from studies WARD Surgery Observational [gov: NCT03491137] and the control group from a WARD Surgery Randomized Controlled Trial (RCT) [gov: NCT04640415 - submitted] were assessed for inclusion eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 691 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
SpO2 <88% in the four hours following opioid administration | four hours following opioid administration

SECONDARY OUTCOMES:
Respiratory deviations four hours after opioid administration | four hours following opioid administration
  SpO2 <92%, <88 %, <85%, <80% and respiratory rate ≤11 min-1, ≤8 min-1, ≤5 min-1

CONTACTS AND LOCATIONS:
Overall Officials: Eske Kvanner Aasvang, Professor, Study Chair — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Bispebjerg Hospital, Copenhagen